CLINICAL TRIAL: NCT04070157
Title: A Randomized, Double-Blind, Placebo-Controlled Pilot Study to Evaluate the Safety and Effectiveness of LUCEMYRA in the Treatment of Opioid Withdrawal During an Opioid Taper in Subjects With Chronic Non-Cancer Pain
Brief Title: Randomized, Double-Blind, Placebo-Controlled Pilot Study on the Safety and Effectiveness of LUCEMYRA During an Opioid Taper in Treatment of Withdrawal
Acronym: TAPER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID pandemic and enrollment issues necessitating an adjustment to the study design.
Sponsor: USWM, LLC (dba US WorldMeds) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USWM-LX1-2010
Record Dates: First submitted 2019-07-02; First posted 2019-08-28 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Opioid Withdrawal (Disorder)
Keywords: Opioid Withdrawal Syndrome; OWS; Opioid taper; Opioid withdrawal; Opioid reduction; Stopping opioids; Opioid discontinuation; non-opioid pain management
MeSH Terms: interventions — lofexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects, study personnel (including the Investigator, study coordinator(s), pharmacist/designee), and the Sponsor will be blinded to the identity of the study drug (active or placebo) administered to subjects.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lofexidine (Experimental)
  Interventions: Drug: Lofexidine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lofexidine — Lofexidine 0.18 mg tablets. Dosing will begin with 1 tablet administered every 5-6 hours, up to 4 times day. The dose may be titrated but not to exceed 4 tablets 4 times a day.
  Other Names: lofexidine hydrochloride; LUCEMYRA
  Arms: Lofexidine
Drug: Placebo — Matching placebo tablets. Dosing will begin with 1 tablet administered every 5-6 hours, up to 4 times day. The dose may be titrated but not to exceed 4 tablets 4 times a day.
  Arms: Placebo

SUMMARY:
Stopping prescription opioid pain medications can be difficult due to withdrawal symptoms. This study will test if LUCEMYRA helps reduce withdrawal symptoms and helps more people reduce their opioid dose compared to placebo.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled pilot study will evaluate the safety and effectiveness of LUCEMYRA in the treatment of opioid withdrawal during an opioid taper in subjects with chronic non-cancer pain.

Subjects will begin a planned 14-day complete taper of their pre-study opioid medications and will be randomly assigned (1:1) to either LUCEMYRA or matching placebo. Study drug will be administered through the opioid taper and for 5 days after the opioid taper is completed. Study drug will then be tapered over a 4-day period for a total of approximately 21 days exposure to study drug.

ELIGIBILITY:
Inclusion Criteria:

* Subject can provide written informed consent.
* Chronic non-cancer pain diagnosis such as low back pain, chronic neck pain, osteoarthritis, and prolonged post-surgical pain with daily pain for a minimum of 6 months.
* Self-reported use of prescribed oral opioid medication(s) (tablets, pills or capsules) of at least 50 morphine mg equivalent (MME) but no higher than 240 mg MME daily or near daily (≥5 days per week) for at least 12 weeks and seeking to discontinue their opioid medication.
* Willing to be treated with non-opioid treatments for pain (in addition to opioid being tapered) for duration of study.
* Willing to abstain from alcohol use during the study.
* Willing to partner with his or her pain physician on a subject-centered pain management plan during the study.
* In generally good health, in the opinion of the Investigator, other than the underlying chronic pain syndrome
* Women of childbearing potential must have a negative pregnancy test at Screening.
* Non-pregnant, non-lactating women who are postmenopausal, naturally or surgically sterile, or who agree to use acceptable contraceptive methods throughout the course of the study.
* Other criteria will be discussed in detail with potential subjects by Site Investigator

Exclusion Criteria:

* Has a primary diagnosis of complex regional pain syndrome, central neuropathic pain, somatoform pain syndromes, acute nerve root compression, any acute or progressive infectious, inflammatory, or neurological process.
* Taking methadone, buprenorphine, fentanyl rapid acting products, tapentadol, tramadol, butorphanol, meperidine, or levorphanol for any reason
* Liver disease that requires medication or medical treatment, and/or AST or ALT levels greater than 3 x ULN.
* Gastrointestinal or renal disease, which would significantly impair absorption, metabolism or excretion of study drug, or would require medication or medical treatment.
* Has a diagnosis of epilepsy or history of seizures.
* Cardiovascular abnormalities at Screening and before randomization (stable hypertension permitted)
* Self-reported or evidence of opioid use disorder (OUD) or other substance use disorder within last 12 months
* Any severe or unstable psychiatric disorder including post-traumatic stress disorder, schizophrenia, bipolar disorder, major depression, substance abuse, or suicidality as determined by the Investigator.
* Subject answers "yes" to "suicidal ideation" in prior 24 months to any items 1 through 5 on the C-SSRS, or subject answers "yes" to any lifetime "suicidal behavior" item on the C-SSRS.
* Any anticipated or scheduled surgery during the study period or within 30 days before Screening.
* Other criteria will be discussed in detail with potential subjects by site Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Peppin, DO, Study Director — US WorldMeds Contract Medical Monitor
Locations (12):
- United States (12):
  - Westview Clinical Research, LLC, Placentia, California
  - Vitamed Research, Rancho Mirage, California
  - Gold Coast Research, LLC, Plantation, Florida
  - Georgia Clinical Research, LLC, Lawrenceville, Georgia
  - Injury Care Research, Boise, Idaho
  - Global Scientific Innovations, Evansville, Indiana
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - Neuroscience Research Center, LLC, Overland Park, Kansas
  - Otrimed Corporation (Otrimed Clinical Research Center), Edgewood, Kentucky
  - University of Rochester, Rochester, New York
  - Duke Innovation Pain Therapies Clinic at Brier Creek, Raleigh, North Carolina
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lofexidine | Placebo
Started | 1 | 3
Completed | 0 | 2
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lofexidine | Placebo | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent AEs and SAEs
Time Frame: Day 1 through Day 28
Measure: Number; unit: participants
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
participants
  Adverse Events | 0 | 5
  Serious Adverse Events | 0 | 0

2. Primary Outcome: Number and Percent of Subjects Reporting TEAEs Resulting in Study Drug Discontinuation
Time Frame: Day 1 through Day 28
Population: There were zero Treatment Emergent AE's.
Measure: Count of Participants; unit: Participants
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
Participants | 0 | 1

3. Primary Outcome: Percentage of Subjects With Treatment-emergent Elevated Liver Function Tests
Time Frame: Day 1 through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
Participants | 0 | 0

4. Primary Outcome: Percentage of Subjects Identified as Suicide Risk With Columbia Suicide Severity Rating Scale
Description: The C-SSRS measures both suicidal ideation and suicidal behavior. The Screener contains "yes" or "no" questions in which respondents are asked to indicate whether they have experienced several thoughts or feelings relating to suicide. A significant risk of suicide is defined as a "yes" in answer to: a) questions 4 or 5 on the suicidal ideation section, or b) any questions on any item in the suicidal behavior section. This must be reported as an SAE and followed up accordingly. Additionally, if a subject responds "yes" to any of the suicidal ideation questions 1 to 3, the Investigator should apply clinical judgment to determine the need for reporting as an AE or SAE and the need for any referral.
Time Frame: Day 1 through Day 28
Population: All responses were "No".
Measure: Number; unit: % of subjects with suicide risk
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
% of subjects with suicide risk | 0 | 0

5. Primary Outcome: Change in Blood Pressure
Description: Orthostatic vital signs were measured in-clinic only. When the subject is at home, only resting vital signs will be collected. Orthostatic vital signs will be measured first after the subject has been sitting for at least 5 minutes and then after the subject has been standing for at least 3 minutes. Resting vital signs only will be measured at home and will be measured after the subject has been sitting quietly for at least 5 minutes.
Time Frame: Baseline to Days 1, 2, 3, 7, 8, 14, 15, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27 and 28
Population: A pause patient in the Placebo group had their End of Study on Visit Day 37. All other participants completed their EOS by Day 28. Orthostatic vital signs only collected in clinic.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Lofexidine: Sitting; Lofexidine: Standing: Lofexidine: Lofexidine 0.18 mg tablets. Dosing will begin with 1 tablet administered every 5-6 hours, up to 4 times day. The dose may be titrated but not to exceed 4 tablets 4 times a day.
- Placebo: Sitting; Placebo: Standing: Placebo: Matching placebo tablets. Dosing will begin with 1 tablet administered every 5-6 hours, up to 4 times day. The dose may be titrated but not to exceed 4 tablets 4 times a day.
Arm/Group | Lofexidine: Sitting | Lofexidine: Standing | Placebo: Sitting | Placebo: Standing
Number analyzed (Participants) | 1 | 1 | 3 | 3
mmHg
  Day 1: Diastolic BP | -2 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.3 (3.06) | -0.7 (3.21)
  Day 1: Systolic BP | -6 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 1.7 (2.31) | -0.3 (1.53)
  Day 2: Diastolic BP: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 2: Diastolic BP | -7 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | 3 (5.66) |
  Day 2: Systolic BP: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 2: Systolic BP | -25 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | 7 (9.9) |
  Day 3: Diastolic BP | -16 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -9 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 1.5 (3.87) | 5 (6)
  Day 3: Systolic BP | -52 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -44 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 6.5 (7.72) | 6 (7.94)
  Day 7: Diastolic BP: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 7: Diastolic BP | -16 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | 7 (8.72) |
  Day 7: Systolic BP: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 7: Systolic BP | -50 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | 6 (7) |
  Day 8: Diastolic BP | -10 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -8 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 3.3 (9.45) | 5.3 (5.86)
  Day 8: Systolic BP | -44 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -36 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 4 (11) | 3 (11)
  Day 14: Diastolic BP: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 14: Diastolic BP | -8 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | 1.7 (10.5) |
  Day 14: Systolic BP: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 14: Systolic BP | -42 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | 4.7 (10.02) |
  Day 15: Diastolic BP | -10 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -4 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 1 (7.81) | 3.3 (7.77)
  Day 15: Systolic BP | -32 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -40 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 10.7 (16.07) | 4.3 (13.01)
  Day 18: Diastolic BP: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 18: Diastolic BP |  |  | 10.7 (6.35) |
  Day 18: Systolic BP: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 18: Systolic BP |  |  | 14.3 (0.58) |
  Day 19: Diastolic BP: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 19: Diastolic BP |  |  | 6.3 (4.5) |
  Day 19: Systolic BP: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 19: Systolic BP |  |  | 11 (6.22) |
  Day 20: Diastolic BP: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 20: Diastolic BP |  |  | 1.8 (5.91) |
  Day 20: Systolic BP: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 20: Systolic BP |  |  | 4.3 (7.68) |
  Day 21: Diastolic BP: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 21: Diastolic BP |  |  | 8.5 (3.42) |
  Day 21: Systolic BP: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 21: Systolic BP |  |  | 11.8 (11.12) |
  Day 22: Diastolic BP | -16 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -8 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 4.3 (3.72) | 10 (1.41)
  Day 22: Systolic BP | -25 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -34 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 9.7 (16.02) | 16 (1.41)
  Day 23: Diastolic BP: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 23: Diastolic BP | -3.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | 3.5 (5.45) |
  Day 23: Systolic BP: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 23: Systolic BP | -19 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | 11.5 (12.23) |
  Day 24: Diastolic BP: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 24: Diastolic BP | -1.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | 6.3 (4.5) |
  Day 24: Systolic BP: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 24: Systolic BP | -23.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | 9.5 (6.61) |
  Day 25: Diastolic BP: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 25: Diastolic BP |  |  | 4.7 (3.56) |
  Day 25: Systolic BP: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 25: Systolic BP |  |  | 8.5 (9.57) |
  Day 26: Diastolic BP: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 26: Diastolic BP | 1.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | 9.3 (7.46) |
  Day 26: Systolic BP: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 26: Systolic BP | -14 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | 8.5 (19.28) |
  Day 27: Diastolic BP: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 27: Diastolic BP |  |  | 4.8 (4.67) |
  Day 27: Systolic BP: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 27: Systolic BP |  |  | 7.7 (8.16) |
  Day 28: Diastolic BP: number analyzed (Participants) | 0 | 0 | 3 | 3
  Day 28: Diastolic BP |  |  | 11 (7.07) | 7.5 (4.95)
  Day 28: Systolic BP: number analyzed (Participants) | 0 | 0 | 3 | 3
  Day 28: Systolic BP |  |  | 22 (7.07) | 15.5 (14.85)
  Day 29: Diastolic BP: number analyzed (Participants) | 0 | 0 | 1 | 0
  Day 29: Diastolic BP |  |  | -0.5 (NA) — No standard deviation because only 1 participant with recorded data. |
  Day 29: Systolic BP: number analyzed (Participants) | 0 | 0 | 1 | 0
  Day 29: Systolic BP |  |  | 18 (NA) — No standard deviation because only 1 participant with recorded data. |
  Day 30: Diastolic BP: number analyzed (Participants) | 0 | 0 | 1 | 0
  Day 30: Diastolic BP |  |  | -1.5 (NA) — No standard deviation because only 1 participant with recorded data. |
  Day 30: Systolic BP: number analyzed (Participants) | 0 | 0 | 1 | 0
  Day 30: Systolic BP |  |  | 8 (NA) — No standard deviation because only 1 participant with recorded data. |
  Day 34: Diastolic BP: number analyzed (Participants) | 0 | 0 | 1 | 0
  Day 34: Diastolic BP |  |  | 0.5 (NA) — No standard deviation because only 1 participant with recorded data. |
  Day 34: Systolic BP: number analyzed (Participants) | 0 | 0 | 1 | 0
  Day 34: Systolic BP |  |  | 12.5 (NA) — No standard deviation because only 1 participant with recorded data. |
  Day 37: Diastolic BP: number analyzed (Participants) | 0 | 0 | 1 | 1
  Day 37: Diastolic BP |  |  | 0 (NA) — No standard deviation because only 1 participant with recorded data. | 3 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 37: Systolic BP: number analyzed (Participants) | 0 | 0 | 1 | 1
  Day 37: Systolic BP |  |  | -5 (NA) — No standard deviation because only 1 participant with recorded data. | -5 (NA) — No standard deviation because only 1 participant with recorded data.

6. Primary Outcome: Change in Pulse
Time Frame: Baseline to Days 1, 2, 3, 7, 8, 14, 15, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27 and 28
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Lofexidine: Sitting | Lofexidine: Standing | Placebo: Sitting | Placebo: Standing
Number analyzed (Participants) | 1 | 1 | 3 | 3
bpm
  Day 1 | 1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -5 (2.65) | -0.3 (3.21)
  Day 2: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 2 | -2 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | -9 (4.24) |
  Day 3 | -4 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -7.3 (2.63) | -5.3 (0.58)
  Day 7: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 7 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | -2 (9.54) |
  Day 8 | -2 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -4 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1 (3.46) | -0.7 (0.58)
  Day 14: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 14 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | -1.7 (7.09) |
  Day 15 | -2 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -11 (8.19) | -3 (3.46)
  Day 18: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 18 |  |  | 1.7 (2.89) |
  Day 19: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 19 |  |  | -2.8 (4.03) |
  Day 20: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 20 |  |  | -8.8 (5.12) |
  Day 21: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 21 |  |  | -1.8 (8.54) |
  Day 22 | -4 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -6 (4.1) | -7 (2.83)
  Day 23: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 23 | 0.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | -4 (11.8) |
  Day 24: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 24 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | -6.5 (4.2) |
  Day 25: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 25 |  |  | -0.8 (7.78) |
  Day 26: number analyzed (Participants) | 1 | 0 | 3 | 0
  Day 26 | 0.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. |  | -9 (4.97) |
  Day 27: number analyzed (Participants) | 0 | 0 | 3 | 0
  Day 27 |  |  | -5.5 (7.31) |
  Day 28: number analyzed (Participants) | 0 | 0 | 3 | 3
  Day 28 |  |  | -7.5 (3.54) | -7 (11.31)
  Day 29: number analyzed (Participants) | 0 | 0 | 1 | 0
  Day 29 |  |  | 3.5 (NA) — Only 1 participant remaining in Placebo group, standard deviation not possible. |
  Day 30: number analyzed (Participants) | 0 | 0 | 1 | 0
  Day 30 |  |  | 1.5 (NA) — Only 1 participant remaining in Placebo group, standard deviation not possible. |
  Day 34: number analyzed (Participants) | 0 | 0 | 1 | 0
  Day 34 |  |  | 2.5 (NA) — Only 1 participant remaining in Placebo group, standard deviation not possible. |
  Day 37: number analyzed (Participants) | 0 | 0 | 1 | 1
  Day 37 |  |  | -13 (NA) — Only 1 participant remaining in Placebo group, standard deviation not possible. | -8 (NA) — Only 1 participant remaining in Placebo group, standard deviation not possible.

7. Secondary Outcome: Percentage of Subjects Who Successfully Complete Each Scheduled Dose Reduction and the Opioid Taper to Complete Opioid Discontinuation
Time Frame: Day 1 through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
Participants | 0 | 2

8. Secondary Outcome: Change in Clinical Opiate Withdrawal Scale (COWS)
Description: The COWS is a clinician-administered instrument that rates 11 common opioid withdrawal signs and symptoms. These include: resting pulse rate; sweating; restlessness; pupil size; bone or joint aches; runny nose or tearing; gastrointestinal upset; tremor; yawning; anxiety or irritability; and gooseflesh skin. Lower total scores indicate a more positive clinical outcome. Score: 5-12 = mild; 13-24 = moderately severe; more than 36 = severe withdrawal. Scores range from a minimum of 0 to a maximum of 48.
Time Frame: Day 1 (pre-1st dose) to Days 3, 8, 15, 22 and 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
score on a scale
  Day 3 | 2 | -0.7 (0.58)
  Day 8 | 3 | -1 (2)
  Day 15 | 4 | -1.3 (0.58)
  Day 22 | -1 | -2.5 (0.71)
  End of Study | -1 | -2.3 (0.58)

9. Secondary Outcome: Change in the Short Opiate Withdrawal Scale of Gossop (SOWS-G)
Description: The SOWS-Gossop scale assesses subjective symptoms of opioid withdrawal. It is a subject-rated scale consisting of 10 items that are scored on a 4-point scale of 0 = none, 1 = mild, 2 = moderate, and 3 = severe (minimum score of 0, maximum score of 30). The overall score is the simple sum of the 10 item scores. Lower observed values in SOWS-Gossop scores indicate a more positive clinical outcome.
Time Frame: Day 1 (pre-1st dose) to Days 1 (at bedtime), 2, 3, 4, 5, 6, 7, 8, 9, 10,11, 12,13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27 and 28
Population: A pause patient in the Placebo group had their End of Study on Visit Day 37. All other participants completed their EOS by Day 28. All remaining blank fields had no data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
score on a scale
  Day 1: number analyzed (Participants) | 0 | 0
  Day 2 | 1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.5 (3)
  Day 3 | 1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -2.2 (3.56)
  Day 4: number analyzed (Participants) | 0 | 3
  Day 4 |  | -0.7 (5.03)
  Day 5 | 1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.3 (5.51)
  Day 6: number analyzed (Participants) | 0 | 3
  Day 6 |  | 0.3 (5.03)
  Day 7 | 1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -2.5 (3.54)
  Day 8 | 1.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.4 (4.72)
  Day 9: number analyzed (Participants) | 0 | 3
  Day 9 |  | 2 (6)
  Day 10 | 4 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -4.5 (0.71)
  Day 11: number analyzed (Participants) | 0 | 3
  Day 11 |  | -0.3 (6.35)
  Day 12 | 2 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -4.5 (0.71)
  Day 13 | 4 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1 (6.08)
  Day 14 | 5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1 (6.08)
  Day 15 | 2.7 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -4.3 (0.96)
  Day 16: number analyzed (Participants) | 0 | 3
  Day 16 |  | 1.5 (6.45)
  Day 17: number analyzed (Participants) | 0 | 3
  Day 17 |  | -4 (1.41)
  Day 18: number analyzed (Participants) | 0 | 3
  Day 18 |  | -4 (1.41)
  Day 19: number analyzed (Participants) | 0 | 3
  Day 19 |  | -4 (1.41)
  Day 20: number analyzed (Participants) | 0 | 3
  Day 20 |  | -4 (1.41)
  Day 21: number analyzed (Participants) | 0 | 3
  Day 21 |  | -4 (1.41)
  Day 22: number analyzed (Participants) | 0 | 3
  Day 22 |  | -3.8 (2.49)
  Day 23: number analyzed (Participants) | 0 | 3
  Day 23 |  | -2.7 (2.52)
  Day 24 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -3 (3)
  Day 25 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -4.5 (2.12)
  Day 26: number analyzed (Participants) | 0 | 3
  Day 26 |  | -3 (3)
  Day 27 | 1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -4 (1.41)
  Day 28: number analyzed (Participants) | 0 | 3
  Day 28 |  | -3.8 (2.87)

10. Secondary Outcome: Change in Subjective Opiate WIthdrawal Scale of Handelsman (SOWS-H)
Description: The SOWS-H scale assesses subjective symptoms of opioid withdrawal. It is a subject-rated scale consisting of 19 items that are scored on a 5-point scale of 0 = not at all, 1 = a little, 2 = moderately, 3 = quite a bit, and 4 = extremely. The overall score is the simple sum of the 19 item scores. Lower observed values in SOWS-H scores indicate a more positive clinical outcome.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
score on a scale
  Day 1: number analyzed (Participants) | 0 | 0
  Day 2 | -4 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0.3 (3.77)
  Day 3 | -5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1 (4.3)
  Day 4: number analyzed (Participants) | 0 | 3
  Day 4 |  | 2.3 (5.51)
  Day 5 | -3 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 3 (6.24)
  Day 6: number analyzed (Participants) | 0 | 3
  Day 6 |  | 3.3 (8.02)
  Day 7 | -4 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0 (5.66)
  Day 8 | -2.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 1.8 (6.3)
  Day 9: number analyzed (Participants) | 0 | 3
  Day 9 |  | 3.5 (7.59)
  Day 10 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.5 (3.54)
  Day 11: number analyzed (Participants) | 0 | 3
  Day 11 |  | 0.7 (6.35)
  Day 12 | -3 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -4 (0)
  Day 13 | 2 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.3 (8.14)
  Day 14 | 1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0.7 (8.96)
  Day 15 | 0.7 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -3.5 (1.29)
  Day 16: number analyzed (Participants) | 0 | 3
  Day 16 |  | 4.3 (9)
  Day 17: number analyzed (Participants) | 0 | 3
  Day 17 |  | -4 (1.41)
  Day 18: number analyzed (Participants) | 0 | 3
  Day 18 |  | -3 (0)
  Day 19: number analyzed (Participants) | 0 | 3
  Day 19 |  | -3 (0)
  Day 20: number analyzed (Participants) | 0 | 3
  Day 20 |  | -3.5 (0.71)
  Day 21: number analyzed (Participants) | 0 | 3
  Day 21 |  | -4 (0)
  Day 22: number analyzed (Participants) | 0 | 3
  Day 22 |  | -2.8 (1.3)
  Day 23: number analyzed (Participants) | 0 | 3
  Day 23 |  | -3.3 (2.08)
  Day 24 | -5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -2.3 (2.89)
  Day 25 | -5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -4.5 (0.71)
  Day 26: number analyzed (Participants) | 0 | 3
  Day 26 |  | -3.3 (2.52)
  Day 27 | -6 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -4 (0)
  Day 28 | -3 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -3.8 (1.89)

11. Secondary Outcome: Modified Clinical Global Impression - Rater Version (MCGI-R) Average Score
Description: MCGI-R includes 2 items: A 7-point scale that allows clinicians to rate the severity of a subject's opiate withdrawal symptoms. A 4-point scale that allows clinicians to rate the degree of a subject's side effects from study drug.
  SEVERITY OF ILLNESS:
  1. = No at all ill
  2. = Borderline ill
  3. = Mildly ill
  4. = Moderately ill
  5. = Markedly ill
  6. = Severely ill
  7. = Among the most extremely ill subjects
  SIDE EFFECTS INDEX:
  1. = None, study drug is producing no side effects
  2. = Do not significantly interfere with subject's functioning
  3. = Significantly interferes with subject's functioning
  4. = Outweighs therapeutic effect
Time Frame: Each scheduled evaluation (Study Visits 2, 3, 4, 5, EOS)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lofexidine Severity of Illness Scale Averages:; Lofexidine Side Effects Index Averages:: Lofexidine: Lofexidine 0.18 mg tablets. Dosing will begin with 1 tablet administered every 5-6 hours, up to 4 times day. The dose may be titrated but not to exceed 4 tablets 4 times a day.
- Placebo Severity of Illness Scale Averages:; Placebo Side Effects Index Averages:: Placebo: Matching placebo tablets. Dosing will begin with 1 tablet administered every 5-6 hours, up to 4 times day. The dose may be titrated but not to exceed 4 tablets 4 times a day.
Arm/Group | Lofexidine Severity of Illness Scale Averages: | Placebo Severity of Illness Scale Averages: | Lofexidine Side Effects Index Averages: | Placebo Side Effects Index Averages:
Number analyzed (Participants) | 1 | 3 | 1 | 3
score on a scale
  Visit 2 | 1 (NA) — Only 1 participant. Standard deviation not possible. | 1 (NA) — Standard deviation not possible as values were the same for all participants. | 1 (NA) — Only 1 participant. Standard deviation not possible. | 1 (NA) — Standard deviation not possible as values were the same for all participants.
  Visit 3 | 1 (NA) — Only 1 participant. Standard deviation not possible. | 1.33 (0.471) | 1 (NA) — Only 1 participant. Standard deviation not possible. | 1.33 (0.471)
  Visit 4 | 1 (NA) — Only 1 participant. Standard deviation not possible. | 1 (NA) — Standard deviation not possible as values were the same for all participants. | 1 (NA) — Only 1 participant. Standard deviation not possible. | 1 (NA) — Standard deviation not possible as values were the same for all participants.
  Visit 5 | 1 (NA) — Only 1 participant. Standard deviation not possible. | 1 (NA) — Standard deviation not possible as values were the same for all participants. | 1 (NA) — Only 1 participant. Standard deviation not possible. | 1 (NA) — Standard deviation not possible as values were the same for all participants.
  EOS | 1 (NA) — Only 1 participant. Standard deviation not possible. | 1 (NA) — Standard deviation not possible as values were the same for all participants. | 1 (NA) — Only 1 participant. Standard deviation not possible. | 1 (NA) — Standard deviation not possible as values were the same for all participants.

12. Secondary Outcome: Modified Clinical Global Impression - Subject Version (MCGI-S)
Description: Includes: A 7-point scale for subjects to rate the severity of opiate withdrawal symptoms. A 4-point scale for subjects to rate the degree of side effects from their study drug.
  SEVERITY OF OPIATE WITHDRAWAL:
  1. = No opiate withdrawal symptoms
  2. = On the border between no to mild opiate withdrawal symptoms
  3. = Mild opiate withdrawal symptoms
  4. = Moderate opiate withdrawal symptoms
  5. = Marked opiate withdrawal symptoms
  6. = Severe opiate withdrawal symptoms
  7. = The most severe opiate withdrawal symptoms that I have ever had
  SIDE EFFECTS INDEX (Scale B):
  1. = None. The study drug has no side effects
  2. = The study drug has slight side effects, but it does NOT significantly interfere with my day to day activities
  3. = The study drug has moderate side effects, and it DOES significantly interfere with my day to day activities
  4. = The study drug has severe side effects, and these side effects are greater than the relief from opiate withdrawal symptoms that it provides
Time Frame: Each scheduled evaluation (Day 1 through Day 28)
Population: No data collection for field with 0 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lofexidine Severity of Opiate Withdrawal Averages:; Lofexidine Side Effects Index Averages:: Lofexidine: Lofexidine 0.18 mg tablets. Dosing will begin with 1 tablet administered every 5-6 hours, up to 4 times day. The dose may be titrated but not to exceed 4 tablets 4 times a day.
- Placebo Severity of Opiate Withdrawal Averages:; Placebo Side Effects Index Averages:: Placebo: Matching placebo tablets. Dosing will begin with 1 tablet administered every 5-6 hours, up to 4 times day. The dose may be titrated but not to exceed 4 tablets 4 times a day.
Arm/Group | Lofexidine Severity of Opiate Withdrawal Averages: | Placebo Severity of Opiate Withdrawal Averages: | Lofexidine Side Effects Index Averages: | Placebo Side Effects Index Averages:
Number analyzed (Participants) | 1 | 3 | 1 | 3
score on a scale
  Day 2 | 1 | 1.33 (0.471) | 1 | 1 (NA) — Standard deviation not possible as values were the same for all participants.
  Day 3 | 1 | 1 (NA) — Standard deviation not possible as values were the same for all participants. | 1 | 1 (NA) — Standard deviation not possible as values were the same for all participants.
  Day 4: number analyzed (Participants) | 0 | 3 | 0 | 3
  Day 4 |  | 2 (NA) — Standard deviation not possible as values were the same for all participants. |  | 2 (NA) — Standard deviation not possible as values were the same for all participants.
  Day 5 | 1 | 1.66 (0.471) | 1 | 1.66 (0.471)
  Day 6: number analyzed (Participants) | 0 | 3 | 0 | 3
  Day 6 |  | 2 (NA) — Standard deviation not possible as values were the same for all participants. |  | 1.66 (0.471)
  Day 7 | 1 | 1.66 (0.471) | 1 | 1.66 (0.471)
  Day 8 | 1 | 2 (NA) — Standard deviation not possible as values were the same for all participants. | 1 | 2 (NA) — Standard deviation not possible as values were the same for all participants.
  Day 9: number analyzed (Participants) | 0 | 3 | 0 | 3
  Day 9 |  | 1.66 (0.471) |  | 1.66 (0.471)
  Day 10 | 1 | 2 (NA) — Standard deviation not possible as values were the same for all participants. | 1 | 1.66 (0.471)
  Day 11: number analyzed (Participants) | 0 | 3 | 0 | 3
  Day 11 |  | 1.66 (0.471) |  | 1.66 (0.471)
  Day 12 | 1 | 2 (NA) — Standard deviation not possible as values were the same for all participants. | 1 | 2 (NA) — Standard deviation not possible as values were the same for all participants.
  Day 13 | 1 | 1.66 (0.471) | 1 | 1.66 (0.471)
  Day 14 | 1 | 2 (NA) — Standard deviation not possible as values were the same for all participants. | 1 | 1.66 (0.471)
  Day 15 | 1 | 1.66 (0.471) | 1 | 1.66 (0.471)
  Day 16: number analyzed (Participants) | 0 | 3 | 0 | 3
  Day 16 |  | 2 (NA) — Standard deviation not possible as values were the same for all participants. |  | 1.66 (0.471)
  Day 17: number analyzed (Participants) | 0 | 2 | 0 | 2
  Day 17 |  | 1.5 (0.5) |  | 1.5 (0.5)
  Day 18: number analyzed (Participants) | 0 | 3 | 0 | 3
  Day 18 |  | 1.5 (0.5) |  | 2 (NA) — Standard deviation not possible as values were the same for all participants.
  Day 19: number analyzed (Participants) | 0 | 2 | 0 | 3
  Day 19 |  | 1.5 (0.5) |  | 2 (NA) — Standard deviation not possible as values were the same for all participants.
  Day 20: number analyzed (Participants) | 0 | 3 | 0 | 3
  Day 20 |  | 1.5 (0.5) |  | 2 (NA) — Standard deviation not possible as values were the same for all participants.
  Day 21: number analyzed (Participants) | 0 | 2 | 0 | 3
  Day 21 |  | 1.5 (0.5) |  | 2 (NA) — Standard deviation not possible as values were the same for all participants.
  Day 22: number analyzed (Participants) | 0 | 3 | 0 | 3
  Day 22 |  | 1.33 (0.471) |  | 1.66 (0.471)
  Day 23: number analyzed (Participants) | 0 | 3 | 0 | 3
  Day 23 |  | 1 (NA) — Standard deviation not possible as values were the same for all participants. |  | 1 (NA) — Standard deviation not possible as values were the same for all participants.
  Day 24 | 1 | 1.33 (0.471) | 1 | 1 (NA) — Standard deviation not possible as values were the same for all participants.
  Day 25: number analyzed (Participants) | 1 | 2 | 1 | 3
  Day 25 | 1 | 1.5 (0.5) | 1 | 1 (NA) — Standard deviation not possible as values were the same for all participants.
  Day 26: number analyzed (Participants) | 0 | 3 | 0 | 3
  Day 26 |  | 1.33 (0.471) |  | 1 (NA) — Standard deviation not possible as values were the same for all participants.
  Day 27: number analyzed (Participants) | 1 | 2 | 1 | 3
  Day 27 | 1 | 1.5 (0.5) | 1 | 1 (NA) — Standard deviation not possible as values were the same for all participants.
  Day 28: number analyzed (Participants) | 0 | 3 | 1 | 3
  Day 28 |  | 1.33 (0.471) | 1 | 1 (NA) — Standard deviation not possible as values were the same for all participants.

13. Secondary Outcome: Time to Study Drug Discontinuation
Description: Study day of participant discontinuation.
Time Frame: Day 1 through Day 28
Measure: Number; unit: Days to study discontinuation
Groups:
- Placebo: Patient 1; Placebo: Patient 2; Placebo: Patient 3: Placebo: Matching placebo tablets. Dosing will begin with 1 tablet administered every 5-6 hours, up to 4 times day. The dose may be titrated but not to exceed 4 tablets 4 times a day.
Arm/Group | Lofexidine | Placebo: Patient 1 | Placebo: Patient 2 | Placebo: Patient 3
Number analyzed (Participants) | 1 | 1 | 1 | 1
Days to study discontinuation | 21 | 20 | 22 | 24

14. Secondary Outcome: Number of Non-opioid Concomitant Medications for Withdrawal Symptoms Used by Study Day
Time Frame: Day 1 through Day 28
Population: No data collection for field with 0 participants.
Measure: Number; unit: Number concomitant medication
Arm/Group | Lofexidine | Placebo: Patient 1 | Placebo: Patient 2 | Placebo: Patient 3
Number analyzed (Participants) | 1 | 1 | 1 | 1
Number concomitant medication
  Day 1-15: | 0 | 1 | 1 | 1
  Day 16- Day 28:: number analyzed (Participants) | 1 | 1 | 1 | 0
  Day 16- Day 28: | 1 | 1 | 1 |

15. Secondary Outcome: Change in EuroQol 5-Dimension 5-Level (EQ-5D-5L) Scale
Description: The EQ-5D-5L is an instrument that evaluates preference for health status through 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each of which are rated on 5 levels of severity. Each dimension ranges from a minimum of "0 - I have no problems or I am not" to a maximum of "5 - I am unable to or I am extremely". The dimensions are averaged together for a single score and the change in average score from baseline is recorded.
Time Frame: Change from Baseline to EOS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
score on a scale | -0.40 (NA) — No standard deviation since only 1 participant analyzed | -0.13 (0.462)

16. Secondary Outcome: Change in Short Form Health Survey (SF-36) Scale
Description: The SF-36 consists of 36 questions that measure various aspects of physical and mental well-being. Precoded values are recorded for each question ranging from 0-100, with a high score defined as a more favorable health status. The items are then averaged together to create the 8 scale scores which are averaged together to create a scale.
  The final value reported is the average change in the averaged scale scores from baseline to end of study.
Time Frame: Change from baseline to End of Study, up to 55 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
score on a scale | -5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.7 (2.52)

17. Secondary Outcome: Change in Insomnia Severity Index (ISI)
Description: The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia. The dimensions evaluated are: severity of sleep onset, sleep maintenance and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item on a scale 0 to 4 for each of the 7 items, yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Time Frame: Change from baseline to Days 15 and End of Study, up to 55 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
score on a scale
  Day 15 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -4 (3)
  EOS | -9 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 1 (1.73)

18. Secondary Outcome: Change in Hospital Anxiety and Depression Scale (HADS)
Description: The HADS is a self-reported screening tool for anxiety and depression in nonpsychiatric clinical populations. Responses are based on the relative frequency of symptoms over the preceding week. The scale consists of 14 items, with a subscale of 7 questions for anxiety and 7 questions for depression. Patients rate each item in the subscales on a 4-point scale ranging from 0 (absence) to 3 (extreme presence). Possible scores range from 0 to 21 for each subscale. An analysis of scores on the 2 subscales supported the differentiation of each mood state into 4 ranges: non-cases (scores 0 to 7), mild cases (scores 8 to 10), moderate cases (scores 11 to 15), and severe cases (scores 16 or higher), with lower values being favorable. The subscales are then combined for a total score ranging from 0 to 42. Higher scores indicate greater levels of anxiety or depression. The value reported is the average change from baseline to End of Study.
Time Frame: Change from End of Study to Baseline, up to 55 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
score on a scale | -2 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -2.3 (3.51)

19. Secondary Outcome: Change in Average Chronic Pain as Measured by the Numeric Rating Scale (NRS)
Description: A subject selects a whole number (0 to 10) that best indicates the intensity of his/her pain.
  The format consists of a horizontal line which is anchored by terms defining pain levels where 0 represents no pain and 10 represents worst pain imaginable.
Time Frame: Baseline through Follow-up (assessed daily)
Population: No data collection for field with 0 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
score on a scale
  Day 1 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.3 (0.82)
  Day 2 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.5 (1)
  Day 3 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.4 (1.82)
  Day 4: number analyzed (Participants) | 0 | 3
  Day 4 |  | -0.7 (1.53)
  Day 5 | -2 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.3 (1.15)
  Day 6: number analyzed (Participants) | 0 | 3
  Day 6 |  | -1 (1)
  Day 7 | -3 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.7 (1.53)
  Day 8 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.8 (2.63)
  Day 9: number analyzed (Participants) | 0 | 3
  Day 9 |  | -1 (0.82)
  Day 10 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.5 (2.12)
  Day 11: number analyzed (Participants) | 0 | 3
  Day 11 |  | -0.3 (1.15)
  Day 12 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1 (2.83)
  Day 13 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1 (2)
  Day 14 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.3 (1.53)
  Day 15 | -0.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.8 (1.5)
  Day 16: number analyzed (Participants) | 0 | 3
  Day 16 |  | -1 (0)
  Day 17: number analyzed (Participants) | 0 | 3
  Day 17 |  | -1 (1.41)
  Day 18: number analyzed (Participants) | 0 | 3
  Day 18 |  | 0 (1.41)
  Day 19: number analyzed (Participants) | 0 | 3
  Day 19 |  | -0.5 (2.12)
  Day 20: number analyzed (Participants) | 0 | 3
  Day 20 |  | 0 (1.41)
  Day 21: number analyzed (Participants) | 0 | 3
  Day 21 |  | -1.5 (2.12)
  Day 22: number analyzed (Participants) | 0 | 3
  Day 22 |  | -1.2 (1.83)
  Day 23: number analyzed (Participants) | 0 | 3
  Day 23 |  | 0 (1.41)
  Day 24 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.7 (1.53)
  Day 25 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.5 (2.12)
  Day 26: number analyzed (Participants) | 0 | 3
  Day 26 |  | -1 (2)
  Day 27 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0 (2.83)
  Day 28: number analyzed (Participants) | 0 | 3
  Day 28 |  | -0.5 (1.73)
  Day 29 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0.7 (1.53)
  Day 30: number analyzed (Participants) | 0 | 3
  Day 30 |  | -0.7 (1.53)
  Day 31 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.7 (1.53)
  Day 32 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.5 (0.71)
  Day 33: number analyzed (Participants) | 0 | 1
  Day 33 |  | -2 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 34: number analyzed (Participants) | 0 | 3
  Day 34 |  | -0.5 (0.71)
  Day 35: number analyzed (Participants) | 0 | 3
  Day 35 |  | -1 (1)
  Day 36: number analyzed (Participants) | 0 | 3
  Day 36 |  | -1 (1.41)
  Day 37 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.8 (0.5)
  Day 38: number analyzed (Participants) | 0 | 3
  Day 38 |  | -1 (1.41)
  Day 39: number analyzed (Participants) | 0 | 3
  Day 39 |  | -1 (1.41)
  Day 40 | 1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.3 (2.08)
  Day 41: number analyzed (Participants) | 0 | 1
  Day 41 |  | -1 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 42: number analyzed (Participants) | 0 | 3
  Day 42 |  | -1 (1.41)
  Day 43 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1 (1.41)
  Day 44: number analyzed (Participants) | 0 | 3
  Day 44 |  | 0 (1.41)
  Day 45 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.5 (0.71)
  Day 46: number analyzed (Participants) | 0 | 3
  Day 46 |  | -0.5 (0.71)
  Day 47 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0 (1.41)
  Day 48 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0 (1.41)
  Day 49: number analyzed (Participants) | 0 | 3
  Day 49 |  | -0.5 (0.71)
  Day 50: number analyzed (Participants) | 0 | 3
  Day 50 |  | -0.5 (0.71)
  Day 51 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0 (1.41)

20. Secondary Outcome: Change in Average Overall Pain as Measured by the Numeric Rating Scale (NRS)
Description: The NRS of pain intensity is a unidimensional, segmented numeric version of the visual analog scale. A subject selects a whole number (0 to 10) that best indicates the intensity of his/her pain. The format consists of a horizontal line which is anchored by terms defining pain levels where 0 represents no pain and 10 represents worst pain imaginable.
Time Frame: Day 1 through Day 28 (assessed daily)
Population: No data collection for field with 0 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
units on a scale
  Day 1 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0 (0)
  Day 2 | -2 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.3 (1.89)
  Day 3 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.4 (2.51)
  Day 4: number analyzed (Participants) | 0 | 3
  Day 4 |  | -0.3 (3.21)
  Day 5 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1 (2.65)
  Day 6: number analyzed (Participants) | 0 | 3
  Day 6 |  | -0.3 (3.21)
  Day 7 | -2 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.7 (2.89)
  Day 8 | -0.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.8 (3.2)
  Day 9: number analyzed (Participants) | 0 | 3
  Day 9 |  | -0.5 (3)
  Day 10 | -2 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -2 (2.83)
  Day 11: number analyzed (Participants) | 0 | 3
  Day 11 |  | -1 (2.65)
  Day 12 | -2 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -2 (2.83)
  Day 13 | -13 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.3 (3.21)
  Day 14 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1 (2.65)
  Day 15 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -2 (2.31)
  Day 16: number analyzed (Participants) | 0 | 3
  Day 16 |  | -0.5 (2.38)
  Day 17: number analyzed (Participants) | 0 | 3
  Day 17 |  | -2 (2.83)
  Day 18: number analyzed (Participants) | 0 | 3
  Day 18 |  | -2 (2.83)
  Day 19: number analyzed (Participants) | 0 | 3
  Day 19 |  | -2 (2.83)
  Day 20: number analyzed (Participants) | 0 | 3
  Day 20 |  | -2 (2.83)
  Day 21: number analyzed (Participants) | 0 | 3
  Day 21 |  | -2 (2.83)
  Day 22: number analyzed (Participants) | 0 | 3
  Day 22 |  | -2 (2.28)
  Day 23: number analyzed (Participants) | 0 | 3
  Day 23 |  | 0 (1.41)
  Day 24 | -2 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.7 (3.06)
  Day 25 | -2 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -2.5 (2.12)
  Day 26: number analyzed (Participants) | 0 | 3
  Day 26 |  | -1.7 (3.06)
  Day 27 | -2 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.5 (0.71)
  Day 28 | 1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.5 (1.91)

21. Secondary Outcome: Change in Worst Chronic Pain as Measured by the Numeric Rating Scale (NRS)
Description: as for outcome 20
Time Frame: Baseline through Day 51 (assessed daily)
Population: No data collection for field with 0 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
score on a scale
  Day 1 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0 (0.63)
  Day 2 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.8 (0.96)
  Day 3 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0.2 (1.3)
  Day 4: number analyzed (Participants) | 0 | 3
  Day 4 |  | 0 (1)
  Day 5 | -3 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0 (1)
  Day 6: number analyzed (Participants) | 0 | 3
  Day 6 |  | 0.7 (0.58)
  Day 7 | -3 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0.3 (0.58)
  Day 8 | -0.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0.3 (0.96)
  Day 9: number analyzed (Participants) | 0 | 3
  Day 9 |  | 0 (0)
  Day 10 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0.5 (0.71)
  Day 11: number analyzed (Participants) | 0 | 3
  Day 11 |  | 1 (1)
  Day 12 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.5 (2.12)
  Day 13 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0.3 (0.58)
  Day 14 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0 (0)
  Day 15 | -0.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0 (0)
  Day 16: number analyzed (Participants) | 0 | 3
  Day 16 |  | 0 (0)
  Day 17: number analyzed (Participants) | 0 | 3
  Day 17 |  | 0 (0)
  Day 18: number analyzed (Participants) | 0 | 3
  Day 18 |  | 1.5 (0.71)
  Day 19: number analyzed (Participants) | 0 | 3
  Day 19 |  | 1.5 (0.71)
  Day 20: number analyzed (Participants) | 0 | 3
  Day 20 |  | 0.5 (0.71)
  Day 21: number analyzed (Participants) | 0 | 3
  Day 21 |  | -1 (1.41)
  Day 22: number analyzed (Participants) | 0 | 3
  Day 22 |  | 0 (0.89)
  Day 23: number analyzed (Participants) | 0 | 3
  Day 23 |  | 0.5 (0.71)
  Day 24 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0.3 (0.58)
  Day 25 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0.5 (0.71)
  Day 26: number analyzed (Participants) | 0 | 3
  Day 26 |  | 0 (1)
  Day 27 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 1.5 (0.71)
  Day 28: number analyzed (Participants) | 0 | 3
  Day 28 |  | 0.5 (0.58)
  Day 29 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 1.3 (0.58)
  Day 30 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0.3 (0.58)
  Day 31 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0.3 (0.58)
  Day 32 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0.5 (0.71)
  Day 33: number analyzed (Participants) | 0 | 1
  Day 33 |  | 1 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 34: number analyzed (Participants) | 0 | 3
  Day 34 |  | 1 (1.41)
  Day 35: number analyzed (Participants) | 0 | 3
  Day 35 |  | 0 (0)
  Day 36: number analyzed (Participants) | 0 | 3
  Day 36 |  | 0 (0)
  Day 37: number analyzed (Participants) | 0 | 3
  Day 37 |  | 0.5 (1)
  Day 38: number analyzed (Participants) | 0 | 3
  Day 38 |  | 0 (0)
  Day 39: number analyzed (Participants) | 0 | 3
  Day 39 |  | 0.5 (0.71)
  Day 40 | 1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0.7 (1.15)
  Day 41: number analyzed (Participants) | 0 | 1
  Day 41 |  | -1 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 42: number analyzed (Participants) | 0 | 3
  Day 42 |  | 0 (0)
  Day 43 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0 (0)
  Day 44: number analyzed (Participants) | 0 | 3
  Day 44 |  | 1.5 (0.71)
  Day 45 | -2 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 1 (1.41)
  Day 46: number analyzed (Participants) | 0 | 3
  Day 46 |  | 1 (1.41)
  Day 47 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 2 (1.41)
  Day 48 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 1 (0)
  Day 49: number analyzed (Participants) | 0 | 3
  Day 49 |  | 0.5 (0.71)
  Day 50: number analyzed (Participants) | 0 | 3
  Day 50 |  | 0.5 (0.71)
  Day 51 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 1 (0)

22. Secondary Outcome: Change in Worst Overall Pain as Measured by the Numeric Rating Scale (NRS)
Description: as for outcome 20
Time Frame: Day 1 through Day 28 (assessed daily)
Population: No data collection for field with 0 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
score on a scale
  Day 1 | 0 (NA) — No standard deviation because only 1 participant in Lofexidine group. | 0 (0)
  Day 2 | -3 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -2.3 (1.53)
  Day 3 | -2.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.6 (1.82)
  Day 4: number analyzed (Participants) | 0 | 3
  Day 4 |  | -0.7 (2.89)
  Day 5 | -3 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1 (1.73)
  Day 6: number analyzed (Participants) | 0 | 3
  Day 6 |  | 0.3 (1.15)
  Day 7 | -2 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1 (2.65)
  Day 8 | 0.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1.8 (2.06)
  Day 9: number analyzed (Participants) | 0 | 3
  Day 9 |  | -0.8 (2.36)
  Day 10 | -4 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -3 (1.41)
  Day 11: number analyzed (Participants) | 0 | 3
  Day 11 |  | -1.7 (2.52)
  Day 12 | -3 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -3 (1.41)
  Day 13 | -2 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -2 (3)
  Day 14 | -1 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -1 (1.73)
  Day 15 | -1.3 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -2.8 (0.96)
  Day 16: number analyzed (Participants) | 0 | 3
  Day 16 |  | -0.8 (2.06)
  Day 17: number analyzed (Participants) | 0 | 3
  Day 17 |  | -3 (1.41)
  Day 18: number analyzed (Participants) | 0 | 3
  Day 18 |  | -2.5 (0.71)
  Day 19: number analyzed (Participants) | 0 | 3
  Day 19 |  | -2.5 (0.71)
  Day 20: number analyzed (Participants) | 0 | 3
  Day 20 |  | -3 (1.41)
  Day 21: number analyzed (Participants) | 0 | 3
  Day 21 |  | -3 (1.41)
  Day 22: number analyzed (Participants) | 0 | 3
  Day 22 |  | -2.7 (1.97)
  Day 23: number analyzed (Participants) | 0 | 3
  Day 23 |  | -1 (2.83)
  Day 24 | -3 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -2 (2.65)
  Day 25 | -3 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -2.5 (0.71)
  Day 26: number analyzed (Participants) | 0 | 3
  Day 26 |  | -2 (2.65)
  Day 27 | -4 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -0.5 (3.54)
  Day 28: number analyzed (Participants) | 0 | 3
  Day 28 |  | -0.5 (1.73)

23. Secondary Outcome: Change in Daily Opioid Dose Expressed as Morphine Equivalent Dose (MED)
Time Frame: Baseline through Day 28
Population: No data collection for field with 0 participants.
Measure: Median (Standard Deviation); unit: MME (morphine milligram equivalent)
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
MME (morphine milligram equivalent)
  Day 1: number analyzed (Participants) | 1 | 1
  Day 1 | -45 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -100 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 2: number analyzed (Participants) | 1 | 1
  Day 2 | -45 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -30 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 3: number analyzed (Participants) | 1 | 2
  Day 3 | -45 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -65 (49.5)
  Day 4 | -45 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -63.3 (35.12)
  Day 5 | -45 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -66.7 (40.41)
  Day 6: number analyzed (Participants) | 0 | 3
  Day 6 |  | -80 (62.45)
  Day 7 | -67.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -75 (25.98)
  Day 8 | -67.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -60.8 (34.13)
  Day 9: number analyzed (Participants) | 0 | 3
  Day 9 |  | -93.3 (50.08)
  Day 10: number analyzed (Participants) | 1 | 2
  Day 10 | -67.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -45 (0)
  Day 11 | -67.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -78.3 (29.3)
  Day 12: number analyzed (Participants) | 1 | 2
  Day 12 | -67.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -67.5 (31.82)
  Day 13: number analyzed (Participants) | 0 | 3
  Day 13 |  | -78.3 (29.3)
  Day 14: number analyzed (Participants) | 0 | 1
  Day 14 |  | -145 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 15: number analyzed (Participants) | 0 | 0
  Day 16: number analyzed (Participants) | 0 | 1
  Day 16 |  | -155 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 17: number analyzed (Participants) | 0 | 0
  Day 18: number analyzed (Participants) | 0 | 0
  Day 19: number analyzed (Participants) | 0 | 0
  Day 20: number analyzed (Participants) | 1 | 0
  Day 20 | -67.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. |
  Day 21: number analyzed (Participants) | 0 | 0
  Day 22: number analyzed (Participants) | 0 | 1
  Day 22 |  | -15 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 23: number analyzed (Participants) | 0 | 1
  Day 23 |  | -20 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 24: number analyzed (Participants) | 1 | 1
  Day 24 | -67.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -20 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 25: number analyzed (Participants) | 1 | 0
  Day 25 | -67.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. |
  Day 26: number analyzed (Participants) | 0 | 0
  Day 27: number analyzed (Participants) | 1 | 0
  Day 27 | -67.5 (NA) — No standard deviation because only 1 participant in Lofexidine group. |
  Day 28: number analyzed (Participants) | 0 | 1
  Day 28 |  | -20 (NA) — No standard deviation because only 1 participant with recorded data.

24. Secondary Outcome: Change in Daily Opioid Dose as a Percentage of the Baseline MED
Time Frame: Baseline through Day 28
Population: No data collection for field with 0 participants.
Measure: Mean (Standard Deviation); unit: MME (morphine milligram equivalent)
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 1 | 3
MME (morphine milligram equivalent)
  Day 1: number analyzed (Participants) | 1 | 1
  Day 1 | -50 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -50 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 2: number analyzed (Participants) | 1 | 1
  Day 2 | -50 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -50 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 3: number analyzed (Participants) | 1 | 2
  Day 3 | -50 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -50 (0)
  Day 4 | -50 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -50 (0)
  Day 5 | -50 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -51.7 (2.89)
  Day 6: number analyzed (Participants) | 0 | 3
  Day 6 |  | -58.3 (14.43)
  Day 7 | -75 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -65 (17.32)
  Day 8 | -75 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -52.1 (21.95)
  Day 9: number analyzed (Participants) | 0 | 3
  Day 9 |  | -74.2 (1.44)
  Day 10: number analyzed (Participants) | 1 | 2
  Day 10 | -75 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -56.3 (26.52)
  Day 11 | -75 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -66.7 (14.43)
  Day 12: number analyzed (Participants) | 1 | 2
  Day 12 | -75 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -75 (0)
  Day 13: number analyzed (Participants) | 0 | 3
  Day 13 |  | -66.7 (14.43)
  Day 14: number analyzed (Participants) | 0 | 1
  Day 14 |  | -72.5 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 15: number analyzed (Participants) | 0 | 0
  Day 16: number analyzed (Participants) | 0 | 1
  Day 16 |  | -77.5 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 17: number analyzed (Participants) | 0 | 0
  Day 18: number analyzed (Participants) | 0 | 0
  Day 19: number analyzed (Participants) | 0 | 0
  Day 20: number analyzed (Participants) | 1 | 0
  Day 20 | -75 (NA) — No standard deviation because only 1 participant in Lofexidine group. |
  Day 21: number analyzed (Participants) | 0 | 0
  Day 22: number analyzed (Participants) | 0 | 1
  Day 22 |  | -7.5 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 23: number analyzed (Participants) | 0 | 1
  Day 23 |  | -10 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 24: number analyzed (Participants) | 1 | 1
  Day 24 | -75 (NA) — No standard deviation because only 1 participant in Lofexidine group. | -10 (NA) — No standard deviation because only 1 participant with recorded data.
  Day 25: number analyzed (Participants) | 1 | 0
  Day 25 | -75 (NA) — No standard deviation because only 1 participant in Lofexidine group. |
  Day 26: number analyzed (Participants) | 0 | 0
  Day 27: number analyzed (Participants) | 1 | 0
  Day 27 | -50 (NA) — No standard deviation because only 1 participant in Lofexidine group. |
  Day 28: number analyzed (Participants) | 0 | 1
  Day 28 |  | -10 (NA) — No standard deviation because only 1 participant with recorded data.

ADVERSE EVENTS:
Time Frame: Day 1 of drug administration through 30 day follow up, up to 57 days.
Arm/Group | Lofexidine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lofexidine (N=1) | Placebo (N=3)
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT04070157/Prot_SAP_002.pdf
  • Informed Consent Form (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT04070157/ICF_001.pdf